CLINICAL TRIAL: NCT05663541
Title: Validity and Reliability of Lower Extremity Position Test in Patients with Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Celal Batuhan Güneysu, Investigator, Pamukkale University
Other Study IDs: E-60116787-020-238650
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis; Sensory Impairments; Proprioceptive Disorders; Validity; Reliability
MeSH Terms: conditions — Multiple Sclerosis; Somatosensory Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient with multiple sclerosis: Patient with multiple sclerosis
  Interventions: Diagnostic Test: Lower extremity position test

INTERVENTIONS:
Diagnostic Test: Lower extremity position test — Assessing proprioception of the lower extremity of individuals multiple sclerosis

SUMMARY:
Sensory disorders are one of the most important problems in individuals with MS, and these disorders are among the first symptoms of MS. Loss of sense of proprioception is particularly common in patients with MS. Studies show that assessment methods for the quantitative measurement of sensory disorders are lacking. Especially in the clinic, there is no evaluation method that evaluates the sense of proprioception. Therefore, the aim of this study perform the validity and reliability study of the lower extremity position test to evaluate proprioception sense in individuals with MS.

ELIGIBILITY:
Inclusion Criteria:

* 20-65 years old
* EDSS score between 0-5
* Person who has not had an attack in the last 1 month or who is not in the attack period
* Person without systemic disease such as hypertension, heart disease, Diabetes Mellitus, hyperlipidemia, malignancy
* Person who has not undergone surgery that restricts balance function in the lower extremity.
* Person without hip, knee and ankle contracture
* Person who does not have additional neurological disease
* Person who does not use vestibulosupressants or drugs that may cause neuropathy and does not have a history of alcohol use
* To have full cooperation and adaptation to the work
* Individuals who agree to receive treatment will be included in the study.

Exclusion Criteria:

* Being younger than 20 years old and over 65 years old
* Being in the attack period
* Hip, knee or ankle contracture
* Being greater than EDSS 5
* Having systemic diseases such as hypertension, heart disease, Diabetes Mellitus, hyperlipidemia, malignancy
* Having an additional neurological disease
* Having a vestibulospressant or drug or alcohol use habit that causes neuropathy
* Not cooperating and adapting to the work

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple sclerosis indivuduals
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Sensorial Assessment-1 | through study completion, an average of 1 year
  Lower Extremity Position test
Sensorial Assessment-2 | through study completion, an average of 1 year
  Kinesthesia (Inclinometer)
Balance Assessment-1 | through study completion, an average of 1 year
  Static Balance via single leg stance
Balance Assessment-2 | through study completion, an average of 1 year
  Dynamic Balance via time up and go
Walking Speed Assessment | through study completion, an average of 1 year
  The 10 meter walk test

SECONDARY OUTCOMES:
Demographic Assessment | through study completion, an average of 1 year
  Demographic form
Expanded Disability Status Scale (EDSS) | through study completion, an average of 1 year
  Ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Romatem Bursa Fizik Tedavi ve Rehabilitasyon Hastanesi, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No